CLINICAL TRIAL: NCT03945929
Title: Can We Alleviate Pain Associated With The Peripheral Intravenous Catheterisation By Using Distraction Methods in Adults: A Randomised Controlled Trial
Brief Title: The Peripheral Intravenous Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Ayla Demirtas, Assistant Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18/7
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researcher, who did not know which patient was in which group, collected the data on the assessment of PIC procedure-associated pain and satisfaction levels immediately after PIC insertion using face-to-face interviews.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Distraction1 group (Experimental): Distraction-1 Group (Cards containing optical illusion pictures)
  Interventions: Behavioral: Distraction
- Control (No Intervention): Control
- Distraction 2 group (Experimental): Distraction-2 Group
  Interventions: Behavioral: Distraction

INTERVENTIONS:
Behavioral: Distraction — Distraction-1 Group: Cards containing approximately six optical illusion pictures were shown to the patients and as a method of distraction during the PIC insertion procedure they were asked what they saw in these cards.
  Distraction-2 Group: Underwater 3D audial videos were played with visual reality (VR) goggles during PIC insertion until the procedure was completed.
  Arms: Distraction 2 group; Distraction1 group

SUMMARY:
Pain management during medical care is considered to be a basic human right and also affects patient satisfaction. In addition, effective management of acute pain contributes to improved patient outcomes. Patient satisfaction is a subjective state that indicates whether the healthcare provided has met the patient's needs and expectations. Many nurse theorists, including Florence Nightingale, have expressed the importance of providing comfort and relief for patients. In fact, comfort has been a crucial aspect of patient care since Nightingale's days, and has been considered an indispensable constituent of integrated nursing care. Studies to improve comfort may contribute to improving individuals' health outcomes, enforcing health-improvement behaviors, and improving healthcare quality as well as satisfaction and contentment of the individual and the nurse in the process of administering healthcare. In the literature, although the efficacy of various pharmacological methods for reducing pain associated with the insertion of PIC has been evaluated in adults, studies on nonpharmacological methods are limited. However, most of the studies were performed in healthy adults. Easy, inexpensive, and fast methods with unlikely side effects are needed to control pain and distress due to the PIC insertion in adults. Therefore, this study was performed to evaluate the effectiveness of distraction methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who ranked 4 (less urgent) and 5 (non-urgent) based on Canadian Emergency Department Triage
* Patients who had no visual, audial, or lingual disabilities, and no mental disorder.

Exclusion Criteria:

* Patients who planned to have PIC insertion and were suitable for having a peripheral intravenous catheter insertion at their antecubital location using 20 Gauge (pink) cannula were eligible.
* Patients who refused to participate in the study,
* Patients who were not eligible for a 20 G peripheral intravenous catheter insertion,
* Patients who could not be inserted a peripheral intravenous catheter at the first time

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Associated With The Peripheral Intravenous Catheterisation | 1-2 minute
  Visual Analog Scale was used to evaluate pain caused by needle insertion. In the Visual Analog Scale of 10 cm length, "0" indicated no pain, and "10" indicated the severest pain.

CONTACTS AND LOCATIONS:
Overall Officials: University of Health Sciences Gulhane Faculty of Nursing, Study Chair — University of Health Sciences Ankara/Turkey
Locations (1):
- Ayla Demirtas, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Basak T, Duman S, Demirtas A. Distraction-based relief of pain associated with peripheral intravenous catheterisation in adults: a randomised controlled trial. J Clin Nurs. 2020 Mar;29(5-6):770-777. doi: 10.1111/jocn.15131. Epub 2019 Dec 16. PMID 31793099

DOCUMENTS (1):
  • Study Protocol (2018-09-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT03945929/Prot_000.pdf